CLINICAL TRIAL: NCT02878395
Title: Genomic/Epigenomic Biomarkers of Deregulation of Immune System in Inflammatory Bowel Diseases: Prediction of Post-operating Natural History of Crohn's Disease
Brief Title: Genomic/Epigenomic Biomarkers of Deregulation of Immune System in Inflammatory Bowel Diseases
Acronym: PREDIPOSTOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PJC 2014/MICI-GERMAIN/MS
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Crohn Disease
Keywords: genomics; epigenomics; recurrence
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ileocolic resection with last loops of small intestine, colon portion and corresponding mesenteric-colic fat.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crohn's disease
  Interventions: Procedure: Ileocolic resection

INTERVENTIONS:
Procedure: Ileocolic resection

SUMMARY:
The purpose is to search for enterocyte-specific or non-specific molecular signature of post-operating recurrence of Crohn's disease in transcriptome (measurement of gene expression through number of mRNA copies transcribed for each gene) and in methylome.

Secondary objectives are to compare expression and methylation profiles according to:

* treatment response
* morphological (endoscopic and/or radiological) and clinical post-operating recurrence.

DETAILED DESCRIPTION:
This aim of this study is to search for new biomarkers predictive of post-operating recurrence.

At present, there are no biomarkers predictive for post-operating recurrence and administration of a post-operating medical treatment to prevent recurrence is based on biological, endoscopic and imagery data.

Predictive biomarkers could allow the identification of patients with high risk of post-operating recurrence and administration of a systematic prophylactic post-operating treatment and at the same time avoiding the prescription of this treatment to patients with low risk of post-operating recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patient with inflammatory bowel disease diagnosis based on clinical (abdominal pain, diarrhea and/or dysenteric syndrome, mostly muco-hemorrhagic, perianal injury, with sometimes general signs and /or systemic manifestations ), biological (inflammatory syndrome, deficiencies…), radiological (entero-MRI), endoscopic (presence of granulomatous lesions) and/or histological (epithelioid and giant cellular granuloma) data
* Patient undergoing ileocolic resection
* Patient affiliated to French social security

Exclusion Criteria:

* Patient refusing sampling
* Patient with undetermined colitis
* Patient with non-confirmed diagnosis of inflammatory bowel disease
* Patient with inflammatory bowel disease not undergoing ileocolic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease needing an ileocolic resection at CHRU Nancy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Gene expression profile in intestinal operative specimens | up to 2 months (from resection)
Methylation profile in intestinal operative specimens | up to 2 months (from resection)

SECONDARY OUTCOMES:
Digestive symptoms | 6, 12, 24 months (after resection)
  such as abdominal pain, Koenig syndrome (abdominal pain relieved by flatus or feces expulsion), diarrhea
Radiological classification of recurrence with entero-MRI performed for post-operating follow-up of patients | 6, 12, 24 months (after resection)
  Koilakou score, recurrence when score >=1
Evaluation of recurrence with endoscopy performed for post-operating follow-up of patients | 6, 12, 24 months (after resection)
  Rutgeerts criteria (recurrence when score >=i1)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline GERMAIN, Principal Investigator — Service de Chirurgie Digestive, Hépatobiliaire, Endocrinienne et Cancérologique CHRU Nancy Brabois Adultes

IPD SHARING:
Plan to Share IPD: No